CLINICAL TRIAL: NCT00634764
Title: Resting Metabolic Rate, Insulin Resistance, and Attitude Towards Weight Gain During Pregnancy to Predict Maternal Weight Gain and Neonatal Body Composition.
Brief Title: Predictors of Maternal Weight Gain and Neonatal Body Composition
Status: Terminated | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Other Study IDs: HR # 16751; GCR Protocol # 769
Record Dates: First submitted 2008-02-19; First posted 2008-03-13 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Obesity
Keywords: Maternal weight gain; Neonatal birth weight; Weight gain attitude; Pregnancy; Body fat; Maternal Behavior; Birth outcomes
MeSH Terms: conditions — Obesity; Gestational Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant: Pregnant women who present to MUSC's Cannon Place or Prenatal Wellness Center

SUMMARY:
Obesity is a significant health issue in the United States with 30% of the US population considered obese defined as a body mass index above 30 kg/m2. Obesity is associated with long term health complications including diabetes and cardiovascular disorders. During pregnancy, obesity is associated with an increased risk of fetal macrosomia and birth injury, as well as increased risk of gestational diabetes, preeclampsia, cesarean birth, and preterm birth. The intrauterine environment has been purported to influence the early childhood and lifelong risk of obesity and the metabolic syndrome (obesity, hyperlipidemia, and insulin resistance [IR]). The Institute of Medicine guidelines for maternal weight gain in pregnancy provide an estimate for population goals, but may be inadequate for individual patient needs. Other factors, such as the degree of maternal IR and resting metabolic rate (RMR) may be more predictive of actual nutritional needs during pregnancy. A better determination of caloric and exercise needs may allow the development of more specific dietary recommendations during pregnancy. Optimal nutrition will result in improved maternal and neonatal outcomes. As the intrauterine environment may have important impacts on neonatal and childhood metabolic and cardiovascular outcomes, creation of a favorable intrauterine environment through optimal maternal nutritional and exercise guidelines may reduce well documented problems such as fetal macrosomia, birth injury, cesarean delivery, and later predisposition toward childhood obesity.

The goal of this pilot trial therefore is to correlate maternal resting metabolic rate, dietary characteristics, and insulin resistance levels with fetal birth weight and body composition in an effort to determine which factors are associated with excessive fat mass in the neonate, placing them at increased lifetime risk of obesity.

We hypothesize that women with lower resting metabolic rates (RMR) in the first trimester will demonstrate a greater maternal weight gain, when adjusted for caloric intake and activity. It is also hypothesized that for a given RMR, the degree of maternal insulin resistance (IR) predicts birthweight adjusted for a given caloric intake. A third hypothesis is that women with increased insulin resistance (measured by HOMA) will result in neonates with larger birth weights and a greater degree of neonatal fat mass as measure by DEXA scan, adjusted for RMR and diet characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Women must be obtaining prenatal care at Cannon Place clinic or at the Prenatal Wellness Center
* Enrolled for prenatal care at less than 16 weeks gestational age
* Singleton pregnancy without fetal abnormalities
* Ability to provide informed consent
* Subjects must complete prenatal visits when data will be collected, and be willing and able to attend three GCRC study visits
* Maternal age >18 and <45
* Neonate born to mother enrolled in trial

Exclusion Criteria:

* Subjects with diabetes, hypertension, prior preterm birth, chronic respiratory disease (asthma on daily medication, COPD, cystic fibrosis) or maternal cardiac disease
* Subjects currently taking insulin sensitizing medications (metformin)
* Subject unable to perform MedGem procedure
* Neonates delivered prior to 34 weeks gestational age will be excluded from analysis by the DEXA scan
* Neonates with fetal anomalies diagnoses in the antenatal period or postpartum will not be included in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of pregnant women who present for prenatal care at MUSC's Cannon Place clinic or Prenatal Wellness Center prior to 16 weeks gestational age.
Sampling Method: Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2006-11 (Actual); Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Maternal weight gain, resting metabolic rate (kcal/day) | During gestation
Neonatal birth weight (gram), ponderal index | After birth

SECONDARY OUTCOMES:
Maternal diet composition, exercise evaluation, insulin resistance, weight gain attitude | During gestation

CONTACTS AND LOCATIONS:
Overall Officials: William Goodnight, MD, Principal Investigator — Medical University of South Carolina; Donna Johnson, Study Chair — Medical University of South Carolina, Obstetrics-Gynecology
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States